CLINICAL TRIAL: NCT03525340
Title: Improving Health Outcomes for HIV-Positive Women in Brazil
Brief Title: Improving Health Outcomes for Women Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 112177; R34MH112177 (NIH)
Record Dates: First submitted 2018-02-28; First posted 2018-05-15 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: HIV/AIDS
Keywords: Engagement to care, peer navigation, transgender
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 2:1 to intervention group with peer navigation or standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants in the standard of care arm will receive no navigation assistance to remain in care. They will provide informed consent, respond to baseline and endline surveys, and have clinic record data extracted for the 9 months of their study participation, but no additional services to remain engaged in care other than what is provided as standard by the clinic.
- Peer Navigation (Experimental): Participants in the peer navigation arm will meet with a peer navigator at least once per month for nine months in-person, and have at least one other navigator contact per month. Like the standard of care arm, they will provide informed consent, respond to baseline and endline surveys, and have clinic record data extracted for the 9 months of their study participation.
  Interventions: Behavioral: Peer Navigation

INTERVENTIONS:
Behavioral: Peer Navigation — Peer navigators help participants identify barriers that pose challenges to the participant's engagement in care and adherence and help develop an overall action plan for addressing these barriers by identifying specific changes that can be made/attempted to overcome an identified barrier. This may involve accompanying a participant to their social services/health appointments, or assisting a participant with disclosure of her HIV status to a family member or friend. The overall goal is to develop knowledge of social/HIV-related health services and good problem-solving skills in order to tackle multiple, potentially overlapping barriers. Over time, participants are encouraged to take increasing degrees of responsibility for identifying and implementing their own problem-solving strategies.
  Arms: Peer Navigation

SUMMARY:
This study will develop and conduct a trans-specific peer navigation intervention in Brazil, which integrates the I-Care approach developed in South Africa with the Model of Gender Affirmation (GA), developed by the investigators to specifically address HIV prevention and care among trans women.

DETAILED DESCRIPTION:
Globally, transgender ('trans') women have 49 times higher odds of HIV infection compared to other groups and trans women living with HIV (TWH) access HIV care and adhere to medication at significantly lower rates than other at-risk groups. Poor engagement in HIV care for TWH is a result of reduced access to and avoidance of healthcare due to stigma and negative experiences with providers, and occurs in the context of social and economic marginalization that foments unstable employment and housing, familial alienation, limited social support, and substance abuse. Interventions to mitigate these barriers to care are critical to reducing HIV-related disparities and poor health outcomes for this highly vulnerable population, particularly where disparities are most apparent, including Brazil. Peer-based navigation (PN) interventions have demonstrated success in improving engagement in HIV care in low-resource settings. The investigators recently conducted a PN intervention ('I-Care') in rural South Africa that significantly improved both linkage to care and retention for men and women. While the PN intervention addresses HIV care engagement by providing social support and skills to work with health providers and family, it requires specific adaptation and a conceptual model that addresses the unique needs of TWH identified during formative research and in consultations with Brazilian stakeholders in 2015. The investigators propose to develop and conduct a trans-specific PN intervention in Brazil, tentatively named 'TransAmigas', which integrates the I-Care approach with the Model of Gender Affirmation (GA), developed by the research team to specifically address HIV prevention and care among trans women. The investigators will use the ADAPT-ITT methodology to develop TransAmigas, incorporating the GA model in the Brazilian context (Aim 1). The investigators will then conduct a pilot study to test the feasibility and acceptability of TransAmigas in São Paulo, Brazil (Aim 2) by randomizing TWH to the intervention (n=100) or to clinical referral (n=50). During the nine month pilot, the investigators will track both navigator and patient adherence to the program, recruitment needs, cohort retention, and reported satisfaction and preferences for program content through surveys at baseline and nine months. Finally, the investigators will prepare for a multi-site efficacy trial (Aim 3) by extracting clinical data from participants' records at the referral clinic, generating preliminary efficacy data by comparing retention in HIV care and viral load by intervention arm. Clinical data will inform future trial sample size. The study will be implemented in Sao Paulo, Brazil, where universal access to care and public support for gender transition care provide an enabling environment for this work to be most effective and where the team has established academic partnerships and a collaboration with the State-run reference and training clinical site (CRT), which includes trans-specific clinical services. If feasible, acceptable, and ultimately proven efficacious, TransAmigas will be the first evidence-based HIV care intervention for TWH globally - filling a crucial gap in programming.

ELIGIBILITY:
Inclusion Criteria:

* have either a recent HIV diagnosis (within the prior 12 months) or be out of care for previously diagnosed HIV
* be a resident of the São Paulo area
* consent for study staff to review their clinical records

Exclusion Criteria:

* female sex at birth
* less than 18 years of age
* not HIV-positive
* currently engaged in care
* unable to provide informed consent
* reside outside of the São Paulo area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male sex at birth, currently identify as female, transgender, transsexual, or travesti (a common term for trans women in Brazil)
Enrollment: 113 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Acceptability of Peer Navigation Intervention | Baseline
  Proportion of transgender women offered navigation services who accept invitation

SECONDARY OUTCOMES:
Feasibility of Peer Navigation Intervention: Patient Satisfaction | At 9 months
  Proportion in TransAmigas who report satisfaction with navigation quality, duration, contact schedule, thematic content, support.
Feasibility of Peer Navigation Intervention: Enrollment rate | At 9 months
  Proportion of transgender women living with HIV who are screened, eligible, enrolled, and successfully complete navigation.
Feasibility of Peer Navigation Intervention: Navigator Retention | At 9 months
  Proportion of navigators who remain in program.
Trial Planning - Linkage to ART | At 9 months
  Time from diagnosis to antiretroviral therapy initiation
Trial Planning - Linkage to confirmatory testing | At 9 months
  Time from diagnosis to CD4+ T-cell count results
Trial Planning - Retention | At 9 months
  Proportion of patients who remain on treatment following 9 months of enrollment in pilot
Trial Planning - Defaulting | At 9 months
  Proportion of participants not in care 90 days after prescribed medication estimated to last 90
Trial Planning - Adherence | At 9 months
  Proportion of days covered (# of dispensed days of medication / # of days between refills)
Trial Planning - Viral Suppression | At 9 months
  Proportion of participants with viral load 1) undetectable and 2) below 1000 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Lippman, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Santa Casa Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Sousa Mascena Veras MA, Menezes NP, Mocello AR, Leddy AM, Saggese GSR, Bassichetto KC, Gilmore HJ, de Carvalho PGC, Maschiao LF, Neilands TB, Sevelius J, Lippman SA. Correlation between gender-based violence and poor treatment outcomes among transgender women living with HIV in Brazil. BMC Public Health. 2024 Mar 13;24(1):791. doi: 10.1186/s12889-024-18224-3. PMID 38481195